CLINICAL TRIAL: NCT06423469
Title: A Multicenter Observational Cohort for the Determination of Noninvasive Intracranial Pressure Waveforms Role in Traumatic Brain Injury
Brief Title: Noninvasive Intracranial Pressure Waveforms Assessment in Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Sergio Brasil, MD (Other)
Collaborators: Braincare USA Corp (Industry)
Responsible Party: Sponsor-Investigator, Sergio Brasil, MD, MD. PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 39348920.1.1001.0068
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; intracranial pressure; intracranial compliance; intracranial pressure waveforms; neurological noninvasive monitoring
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TBI patients: TBI patients to be monitored daily with the brain4care system for fifteen days
  Interventions: Device: Noninvasive ICP monitoring

INTERVENTIONS:
Device: Noninvasive ICP monitoring — The brain4care system is a FDA approved noninvasive device for surrogate intracranial pressure monitoring. Serial monitoring sessions were performed in included patients. Information recorded was for study purposes only and did not affect any therapy planned for the attending teams.

SUMMARY:
In clinical practice, hospital admission of patients with altered level of consciousness ranging from drowsiness to decreasing response states or coma is extremely common. This clinical condition demands effective investigation and early treatment. Imaging and laboratory tests have played increasingly relevant roles in supporting clinical research. One of the main causes of coma is intracranial hypertension (IH), with traumatic brain injuries (TBI) and cerebral hemorrhages being the major contributors to its development. IH increases the risk of secondary damage in these populations, and consequently, morbidity and mortality. Clinical studies show that adequate intracranial pressure (ICP) control in TBI patients reduces mortality and increases functionality. Unfortunately, the most accurate way to measure and evaluate the ICP is through a catheter located inside the skull, and its perforation is required for this purpose. Several studies have attempted to identify noninvasive solutions for ICP monitoring; however, to date, none of the techniques gathered sufficient evidence to replace invasive monitors. Recently, an extensometer device has been developed, which only maintains contact with the skull's skin and therefore eliminates the need for its perforation, being able to obtain recordings of cranial dilatation at each heartbeat and consequently reflecting brain compliance. In vivo studies have identified excellent qualitative correlation with catheter ICP recordings. However, this device was evaluated only in a limited number of clinical cohorts and the correlations between the information provided by this device with patients outcomes is still poor. Therefore, this project aims primarily to evaluate the use of this noninvasive brain compliance monitoring system in a cohort of TBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe traumatic brain injury with less than 24 hours.

Exclusion Criteria:

* Primary decompressive craniectomy
* Brain death signs at admission
* Severe hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of any gender, older than 18 years, with very acute moderate or severe TBI will be included just after stabilization and any surgical evacuation procedure performed.
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | One month
  Is in-hospital mortality correlated with poorer brain4care biometrics?

SECONDARY OUTCOMES:
Morbidity | Six months
  Is morbidity correlated with poorer brain4care biometrics?

OTHER OUTCOMES:
Correlation with invasive information | Fifteen days
  Are brain4care biometrics correlated with invasive intracranial pressure provided by ventricular catheters or parenchymal probes?

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Universidade Federal do Amazonas, Manaus, Amazonas
  - Hospital João XXIII, Belo Horizonte, Minas Gerais
  - Hospital de Emergência e Trauma Senador Humberto Lucena, João Pessoa, Paraíba
  - Universidade de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
Possibly some anonymous data can be shared with other researchers upon reasonable request.

REFERENCES:
- [Background] Gulamali F, Jayaraman P, Sawant AS, Desman J, Fox B, Chang A, Soong BY, Arivazaghan N, Reynolds AS, Duong SQ, Vaid A, Kovatch P, Freeman R, Hofer IS, Sakhuja A, Dangayach NS, Reich DS, Charney AW, Nadkarni GN. Derivation, External Validation and Clinical Implications of a deep learning approach for intracranial pressure estimation using non-cranial waveform measurements. medRxiv [Preprint]. 2024 Jan 30:2024.01.30.24301974. doi: 10.1101/2024.01.30.24301974. PMID 38352556
- [Background] Kawoos U, McCarron RM, Auker CR, Chavko M. Advances in Intracranial Pressure Monitoring and Its Significance in Managing Traumatic Brain Injury. Int J Mol Sci. 2015 Dec 4;16(12):28979-97. doi: 10.3390/ijms161226146. PMID 26690122
- [Background] de Moraes FM, Rocha E, Barros FCD, Freitas FGR, Miranda M, Valiente RA, de Andrade JBC, Neto FEAC, Silva GS. Waveform Morphology as a Surrogate for ICP Monitoring: A Comparison Between an Invasive and a Noninvasive Method. Neurocrit Care. 2022 Aug;37(1):219-227. doi: 10.1007/s12028-022-01477-4. Epub 2022 Mar 24. PMID 35332426
- [Background] de Moraes FM, Brasil S, Frigieri G, Robba C, Paiva W, Silva GS. ICP wave morphology as a screening test to exclude intracranial hypertension in brain-injured patients: a non-invasive perspective. J Clin Monit Comput. 2024 Aug;38(4):773-782. doi: 10.1007/s10877-023-01120-3. Epub 2024 Feb 14. PMID 38355918
- [Background] Brasil S, Solla DJF, Nogueira RC, Teixeira MJ, Malbouisson LMS, Paiva WDS. A Novel Noninvasive Technique for Intracranial Pressure Waveform Monitoring in Critical Care. J Pers Med. 2021 Dec 5;11(12):1302. doi: 10.3390/jpm11121302. PMID 34945774